CLINICAL TRIAL: NCT00946842
Title: A Phase I, Two-Panel, Open-Label, Randomized, 3-way Crossover Trial in Healthy Subjects to Determine the Relative Oral Bioavailability of TMC207 After Single Dose Administration of TMC207 100 mg as the Phase II Clinical Trial Tablet Formulation and as a Newly Developed Tablet Formulation, Under Fed and Fasted Conditions
Brief Title: A Study to Determine the Relative Oral Bioavailability of Single Dose Administration of TMC207, Under Fed and Fasted Conditions in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR007504; TMC207-TIDP13-C111 (Other: Tibotec-Virco Virology BVBA); TMC207-C111 (Other: Tibotec-Virco Virology BVBA)
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Healthy; Bioavailability; Relative bioavailability; TMC207; Fed condition; Fasted condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Panel A: Treatment Sequence ABC (Experimental): Participants will receive the 3 treatments (Treatment A,B and C) in sequence ABC with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel A: Treatment Sequence ACB (Experimental): Participants will receive the 3 treatments (Treatment A,B and C) in sequence ACB with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel A: Treatment Sequence BAC (Experimental): Participants will receive the 3 treatments (Treatment A,B and C) in sequence BAC with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel A: Treatment Sequence BCA (Experimental): Participants will receive the 3 treatments (Treatment A,B and C) in sequence BCA with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel A: Treatment Sequence CBA (Experimental): Participants will receive the 3 treatments (Treatment A,B and C) in sequence CBA with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel A: Treatment Sequence CAB (Experimental): Participants will receive the 3 treatments (Treatment A,B and C) in sequence CAB with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel B: Treatment Sequence DEF (Experimental): Participants will receive the 3 treatments (Treatment D,E and F) in sequence DEF with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel B: Treatment Sequence DFE (Experimental): Participants will receive the 3 treatments (Treatment D,E and F) in sequence DFE with food and subsequent treatments will be separated by 4 weeks..
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel B: Treatment Sequence EDF (Experimental): Participants will receive the 3 treatments (Treatment D,E and F) in sequence EDF with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel B: Treatment Sequence EFD (Experimental): Participants will receive the 3 treatments (Treatment D,E and F) in sequence EFD with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel B: Treatment Sequence FDE (Experimental): Participants will receive the 3 treatments (Treatment D,E and F) in sequence FDE with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel B: Treatment Sequence FED (Experimental): Participants will receive the 3 treatments (Treatment D,E and F) in sequence FED with food and subsequent treatments will be separated by 4 weeks.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F

INTERVENTIONS:
Drug: Treatment A — Participants will receive phase II clinical study tablet formulation of TMC207 100 mg as a single oral dose with food on Day 1, Day 30 and Day 58.
  Arms: Panel A: Treatment Sequence ABC; Panel A: Treatment Sequence ACB; Panel A: Treatment Sequence BAC; Panel A: Treatment Sequence BCA; Panel A: Treatment Sequence CAB; Panel A: Treatment Sequence CBA
Drug: Treatment B — Participants will receive newly developed tablet formulation with fine particle size distribution of TMC207 100 mg as a single oral dose with food on Day 1, Day 30 and Day 58.
  Arms: Panel A: Treatment Sequence ABC; Panel A: Treatment Sequence ACB; Panel A: Treatment Sequence BAC; Panel A: Treatment Sequence BCA; Panel A: Treatment Sequence CAB; Panel A: Treatment Sequence CBA
Drug: Treatment C — Participants will receive newly developed tablet formulation with coarse particle size distribution of TMC207 100 mg as a single oral dose with food on Day 1, Day 30 and Day 58.
  Arms: Panel A: Treatment Sequence ABC; Panel A: Treatment Sequence ACB; Panel A: Treatment Sequence BAC; Panel A: Treatment Sequence BCA; Panel A: Treatment Sequence CAB; Panel A: Treatment Sequence CBA
Drug: Treatment D — Participants will receive phase II clinical study tablet formulation of TMC207 100 mg as a single oral dose without food on Day 1, Day 30 and Day 58.
  Arms: Panel B: Treatment Sequence DEF; Panel B: Treatment Sequence DFE; Panel B: Treatment Sequence EDF; Panel B: Treatment Sequence EFD; Panel B: Treatment Sequence FDE; Panel B: Treatment Sequence FED
Drug: Treatment E — Participants will receive newly developed tablet formulation with fine particle size distribution of TMC207 100 mg as a single oral dose without food on Day 1, Day 30 and Day 58.
  Arms: Panel B: Treatment Sequence DEF; Panel B: Treatment Sequence DFE; Panel B: Treatment Sequence EDF; Panel B: Treatment Sequence EFD; Panel B: Treatment Sequence FDE; Panel B: Treatment Sequence FED
Drug: Treatment F — Participants will receive newly developed tablet formulation with coarse particle size distribution of TMC207 100 mg as a single oral dose without food on Day 1, Day 30 and Day 58
  Arms: Panel B: Treatment Sequence DEF; Panel B: Treatment Sequence DFE; Panel B: Treatment Sequence EDF; Panel B: Treatment Sequence EFD; Panel B: Treatment Sequence FDE; Panel B: Treatment Sequence FED

SUMMARY:
The purpose of this study is to determine the relative oral bioavailability (the extent to which a medication or other substance becomes available to the body as compared with another form of medication or other substance) of TMC207 after single-dose oral administration of the Phase II clinical study tablet formulation, and a newly developed tablet formulations, under fed (with food) and fasted (without food) conditions.

DETAILED DESCRIPTION:
This is a 2-panel (2 groups), open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), 3- way crossover (method used to switch participants from one treatment arm to another in a clinical study) study. The study consists of 3 phases including, the screening phase (less than or equal to 21 days before administration of study medication), treatment phase (84 days), and the follow-up phase (up to 30 to 35 days after the last blood sample in the last treatment session is collected). Approximately 24 healthy participants will be allocated to one of two panels: Panel A (participants will receive study medication under fed condition); and Panel B (participants will receive study medication under fasted condition). Participants in Panel A will be randomly assigned to 1 of 6 treatment sequences (Treatment sequences ABC, ACB, BAC, BCA, CBA, and CAB) to receive the following 3 formulations of TMC207 with food: Treatments A: the Phase II tablet formulation; Treatment B: newly developed tablet formulation with fine particle size distribution; and Treatment C: newly developed tablet formulation with coarse particle size distribution. Participants in Panel B will be randomly assigned to 1 of 6 treatment sequences (Treatment sequences DEF, DFE, EDF, EFD, FDE, and FED) to receive the following 3 formulations of TMC207 without food: Treatments D: the Phase II tablet formulation; Treatment E: newly developed tablet formulation with fine particle size distribution; and Treatment F: newly developed tablet formulation with coarse particle size distribution. Subsequent treatments will be separated by a period of 4 weeks. The total duration of the study for each participant will be approximately 20 weeks. Safety evaluations will include assessment of adverse events, clinical laboratory tests, vital signs, electrocardiogram, physical examination, and alcohol urine medicine screen which will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker or smokers with no more than 10 cigarettes or 2 cigars or 2 pipes per day for at least 3 months prior selection
* Normal weight as defined by a body mass index (weight in kilograms divided by the square of height in meters) of 18 to 30 kg/m2, extremes included
* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality

Exclusion Criteria:

* Positive tests for Human Immunodeficiency Virus 1 (HIV type 1) or HIV 2; hepatitis A, hepatitis B, or hepatitis C infection; and urine drug tests at screening
* Female with no childbearing potential
* History or current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use
* Relevant medical history or presence of systemic disease (gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, infectious disease), or significant skin disease
* History or presence of clinically significant electrocardiogram at screening
* Abnormal laboratory values at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Time to Reach the Maximum Plasma Concentration of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Maximum Plasma Concentration of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Area Under Curve From Time of Administration up to 72 Hours Post Dosing of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration

SECONDARY OUTCOMES:
Time to Reach the Maximum Plasma Concentration of M2 Metabolite of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Maximum Plasma Concentration of M2 Metabolite of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Area Under Curve From Time of Administration up to 72 Hours Post Dosing of M2 Metabolite of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Area Under Curve From Time of Administration up to the Last Time Point With a Measurable Concentration Post Dosing of M2 Metabolite of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Area Under Curve Extrapolated to Infinity of M2 Metabolite of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Elimination Rate Constant of a Sequential Elimination Phase of the Plasma Concentration-Time Curve of M2 Metabolite of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Elimination Half-Life of M2 Metabolite of TMC207 | 0 hour predose to 672 hours postdose, after each of the 3 single-dose administration
Number of Participants With Adverse Events | Up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA